CLINICAL TRIAL: NCT06506045
Title: Measurements of Flow in Functional and Non-Functional Cerebrospinal Fluid Shunts With a Second-Generation Wireless Thermal Anisotropy Measurement Device
Brief Title: Functional and Non-Functional CSF Shunt Flow Measured With a Second-Generation Wireless Thermal Device
Status: Terminated | Type: Observational
Why Stopped: Enrollment
Sponsor: Rhaeos, Inc. (Industry)
Responsible Party: Sponsor
Other Study IDs: 2024-02
Record Dates: First submitted 2024-07-11; First posted 2024-07-17 (Actual); Last update posted 2025-05-15 (Actual); Status verified 2025-05

CONDITIONS: Hydrocephalus
MeSH Terms: conditions — Hydrocephalus

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: No

INTERVENTIONS:
Device: FlowSense — This study compares the performance of two generations of non-invasive cerebrospinal fluid (CSF) shunt flow assessment devices. Measurements of known non-functional and functional implanted shunts will assess the diagnostic non-inferiority of the second-generation device to the first-generation device.

SUMMARY:
This study compares the performance of two generations of non-invasive cerebrospinal fluid (CSF) shunt flow assessment devices. Measurements of known non-functional and functional implanted shunts will assess the diagnostic non-inferiority of the second-generation device to the first-generation device.

ELIGIBILITY:
Inclusion Criteria:

1. At least one existing ventricular CSF shunt, functional or non-functional (including an adjustable valve set to "virtual off," ligated shunt, uncorrected distal catheter disconnection or fracture, distal catheter fragment left in place during shunt surgery, or indication that the shunt is otherwise non-functional), with a region of overlying intact skin appropriate in size for application of the study device
2. If more than one distal shunt catheter is present, at least one distal shunt catheter is at least 2 cm away from any other distal shunt catheter in the device measurement region
3. Signed informed consent by subject or a parent, legal guardian, health care agent, or surrogate decision maker (according to local statutes)
4. Signed medical records release by subject or a parent, legal guardian, health care agent, or surrogate decision maker (according to local statutes)
5. Verbal assent by minors 7 years of age and older who are able to understand the study and communicate their decision

Exclusion Criteria:

1. Presence of an interfering open wound or edema in the FlowSense device measurement area
2. Patient-reported history of adverse skin reactions to adhesives
3. Previous participation in a Rhaeos clinical study in which FlowSense device measurement data were acquired
4. New or worsening symptoms of a possible shunt malfunction in the prior 7 days
5. Use of the study device would interfere with standard patient care, or emergency surgery that cannot be delayed, or participation in the study will interfere with, or be detrimental to, administration of optimal healthcare to the subject
6. Participation in any other investigational procedural, pharmaceutical, and/or device study that may influence the collection of valid data under this study

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Pediatric and adult patients with an existing ventricular shunt will be enrolled in this study.
Sampling Method: Non-Probability Sample
Enrollment: 10 (Actual)
Dates: Start 2024-07-27 (Actual); Primary Completion 2024-07-27 (Actual); Study Completion 2024-07-27 (Actual)

PRIMARY OUTCOMES:
Study Device Sensitivity | Up to 1 hour
  Study device sensitivity will be calculated as TP / (TP + FN).
Study Device Specificity | Up to 1 hour
  Study device specificity will be calculated as TN / (TN + FP)

CONTACTS AND LOCATIONS:
Locations (8):
- United States (8):
  - CHOC Commerce Tower, Orange, California
  - Cedars-Sinai Accelerator, West Hollywood, California
  - Tampa Marriott Water Street, Tampa, Florida
  - MATTER, Chicago, Illinois
  - Industrious, Evanston, Illinois
  - Northwest Special Recreation Association, Rolling Meadows, Illinois
  - Texas Medical Center Innovation, Houston, Texas
  - Industrious, Seattle, Washington